CLINICAL TRIAL: NCT06765499
Title: A Prospective, Double-blind, Randomized Controlled Study Evaluating the Improvement of Nutritional Status and Frailty With Silkworm Pupa Powder Compared With Placebo Among Motor Neuron Disease
Brief Title: The Study Evaluating the Improvement of Nutritional Status and Frailty With Silkworm Pupa Powder Among Patients With Motor Neuron Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First People's Hospital of Hangzhou (Other)
Collaborators: Hangzhou Institute of Medicine Chinese Academy of Sciences (Unknown)
Responsible Party: Principal Investigator, Buqing Ma, M.M., Associate Director of Motor Neuron Disease piagnosis and Treatment center, First People's Hospital of Hangzhou
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZN-2024308-02
Record Dates: First submitted 2024-12-11; First posted 2025-01-09 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-01

CONDITIONS: Motor Neuron Disease (MND); Amyotrophic Lateral Sclerosis (ALS)
Keywords: Amyotrophic Lateral Sclerosis; Motor Neuron Disease; Frailty; Nutritional Status
MeSH Terms: conditions — Motor Neuron Disease; Amyotrophic Lateral Sclerosis; Frailty

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Silkworm pupa powder (Experimental): The intervention in the trial involves providing silkworm pupa powder, twice a day, with two packets each time, to be taken before meals.The dose of gastrointestinal weak people was halved, twice a day, 1 pack each time, half an hour before breakfast and dinner.
  Interventions: Other: Chinese medicine - Silkworm pupa powder
- Placebo (Placebo Comparator): The intervention for the placebo group involves administering a placebo containing 0.5% of the active ingredient, twice daily, with two packets each time, taken before meals.The dose of gastrointestinal weak people was halved, twice a day, 1 pack each time, half an hour before breakfast and dinner.
  Interventions: Other: Ultra-low dose silkworm pupa powder

INTERVENTIONS:
Other: Chinese medicine - Silkworm pupa powder — Silkworm pupa contains high-quality animal protein and has a wide range of activities in antioxidant, antitumor, antibacterial, and immune enhancement, making it highly nutritious and medicinally valuable.
  Arms: Silkworm pupa powder
Other: Ultra-low dose silkworm pupa powder — 0.5% of the effective components in the experimental group
  Arms: Placebo

SUMMARY:
Motor Neuron Disease (MND) is the result of dysfunction of the upper motor neurons in the precentral gyrus of the frontal lobe or the lower motor neurons in the ventral horn of the spinal cord. Amyotrophic lateral sclerosis (ALS) is the most common, disabling, and fatal motor neuron disease in adults. Sarcopenia is a syndrome characterized by progressive loss of skeletal muscle mass, accompanied by a reduction in muscle strength and (or) function, and it is an important feature of MND. Aging is an objective and inevitable process that involves the gradual degeneration and loss of physiological functions in various tissues, organs, and cells. With the continuous accumulation of various injuries, the body eventually exhibits signs of frailty such as fatigue, reduced muscle strength, and weight loss. Data from adult ALS patients indicate that 58% of patients are at risk of frailty. Silkworm pupa contains high-quality animal protein and has a wide range of activities in antioxidant, antitumor, antibacterial, and immune enhancement, making it highly nutritious and medicinally valuable. Silkworm pupa extracts can enhance grip strength in older adults with relatively low skeletal muscle mass. As a natural food ingredient with high safety, the value of silkworm pupa in ALS patients lacks corresponding research, which limits its further application in clinical practice. This study aims to select ALS patients as the research subjects and use a randomized, controlled, double-blind prospective study design to evaluate the effectiveness of silkworm pupa tablets in improving sarcopenia, frailty, and quality of life in ALS patients. The study strives to improve the frailty condition of ALS patients and enhance their quality of life by supplementing nutrition, thereby providing new strategies for comprehensive intervention and management of ALS patients.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participate in the clinical study, fully understand and be informed about the study, and sign the Informed Consent Form (ICF); willing to follow and capable of completing all trial procedures.
* Gender is not limited, age at the time of signing ICF: ≥18 years old, ≤80 years old; if the ALS patient is at least 18 years old, then the weight must be over 40 kilograms.
* Diagnosis conforms to the confirmed and probable ALS in the ALS2020 diagnostic criteria (Gold Coast Criteria).
* Clinical, neurophysiological, or pathological examination confirms evidence of lower motor neuron involvement.
* Frailty Phenotype scale (FP) ≥1.
* Exclude other diseases.
* Agree to provide peripheral blood, fecal, and urine samples for biomarker analysis during the study period.

Exclusion Criteria:

* Patients with other neurological diseases similar to ALS symptoms or affecting drug efficacy evaluation, such as cervical spondylosis, lumbar disease, dementia, etc.
* Patients with other autoimmune diseases, such as Multiple Sclerosis (MS), Polymyositis, Myasthenia Gravis, Guillain-Barré Syndrome, Ankylosing Spondylitis, Rheumatoid Arthritis, Systemic Lupus Erythematosus, Vitiligo, etc.
* Severe renal insufficiency: Creatinine clearance < 30 mL/min (Cockcroft-Gault formula), or other known severe renal insufficiency diseases.
* Severe liver damage: ALT, AST > 3 times the upper limit of normal, or other known liver diseases such as acute and chronic active hepatitis, cirrhosis, etc.
* Patients with severe pulmonary function insufficiency such as Chronic Obstructive Pulmonary Disease (COPD), pulmonary fibrosis, etc.
* During the screening period, patients with acute myocardial infarction or interventional treatment within the last 6 months, heart failure patients (classified as NYHA class III-IV patients).
* Patients with other severe primary diseases of the nervous system, heart, lungs, hematopoietic system, or endocrine system, and mental illness patients.
* Those suspected or confirmed to have a history of alcohol or drug abuse.
* Expected survival ≤ 3 months.
* Pregnant or breastfeeding women, subjects of reproductive age (including male subjects who have had heterosexual intercourse and their female partners with childbearing potential) who plan to become pregnant or are unwilling to take effective contraceptive measures from the start of screening to 3 months after discontinuing medication.
* Those who are allergic to known ingredients of the trial products; or have a history of drug allergies or severe allergic diseases (anaphylactic shock, etc.).
* During the study, individuals assessed by researchers as potential drug abusers who may affect the efficacy of therapeutic drugs.
* Presence of other severe physical or mental diseases or abnormal laboratory tests that may increase the risk of participating in the study and patients deemed unsuitable for participation by the researcher.
* Patients with malignant tumors.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Assessing patient nutritional improvement using Third Lumbar Skeletal Muscle Index (L3-SMI). | The 0th、 4th 、8th and 12th week after taking Silkworm Silkworm pupa powder.
  The nutritional index is evaluated using the Third Lumbar Skeletal Muscle Index (L3-SMI): A single cross-sectional image of L3 is obtained through CT scanning, and skeletal muscles in the image are identified and quantified using a HU threshold of -29 to 150. The total muscle area at this level is calculated using 3D Slicer software, and then divided by the square of the height (m^2) to obtain the Third Lumbar Skeletal Muscle Index (L3-SMI).
The improvement of frailty in patients treated by the Frailty Phenotype (FP) Scale assessment. | The 0th、 4th 、8th and 12th week after taking Silkworm Silkworm pupa powder.
  Frailty Phenotype Scale: The Frailty Phenotype (FP) Scale encompasses the following five clinical criteria:
  * Unintentional Weight Loss
  * Self-reported Fatigue
  * Decreased Physical Activity
  * Slowed Gait Speed
  * Weak Grip Strength Each criterion is scored as 1 point if met, with a total score ranging from 0 to 5. A score of 0 indicates robust health, a score of 1 to 2 indicates pre-frailty, and a score of 3 or higher indicates frailty.
  This scale is used to assess the frailty status of individuals, providing a separate outcome measure that focuses on the physical vulnerability and decreased resilience commonly associated with aging.

SECONDARY OUTCOMES:
Using the Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R) to assess patient functional status, thereby evaluating the improvement of neurological dysfunction. | The 0th、 4th 、8th and 12th week after taking Silkworm Silkworm pupa powder.
  Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R) consists of 12 items with a total score of 48 points, where each item is rated from 0 to 4, with 0 indicating complete loss of function and 4 indicating normal function.
  The minimum score is 0 points, which indicates that the patient is completely unable to perform any of the tasks listed in the scale, while the maximum score is 48 points, indicating that the patient can perform all tasks normally.
  A higher score implies better functional status in the patient, meaning less severe neurological impairment; a lower score indicates worse functional status, meaning more severe neurological impairment.
  This scale is a specific tool for evaluating the functional status of patients with Amyotrophic Lateral Sclerosis, offering a distinct outcome measure that quantifies the progression of the disease.
Assess the respiratory function of patients with Amyotrophic Lateral Sclerosis undergoing treatment using the Oxygenation Index. | The 0th、 4th 、8th and 12th week after taking Silkworm Silkworm pupa powder.
  Oxygenation Index: The Oxygenation Index combines arterial oxygen partial pressure (PaO2) and inspired oxygen fraction (FiO2), calculated using the formula Oxygenation Index (mmHg) = PaO2 (mmHg) / FiO2 (%). It provides a single value indicating a patient's oxygenation status relative to the oxygen concentration they are breathing, thereby characterizing respiratory function. During the treatment process, the change coefficients of the Oxygenation Index after intervention in the silkworm pupa treatment group and the placebo group are calculated, using this coefficient to characterize the relief ratio of respiratory function following Silkworm pupa powder intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Hangzhou First People's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No